CLINICAL TRIAL: NCT06767956
Title: Phase I/II Study of Combination Golcadomide and Nivolumab in Patients With Non-Hodgkin Lymphoma With Refractory Disease After Chimeric Antigen T-cell Therapy
Brief Title: Golcadomide and Nivolumab in Patients With Non-Hodgkin Lymphoma With Refractory Disease After Chimeric Antigen T-cell Therapy
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Natalie Galanina (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Natalie Galanina, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 23-161
Record Dates: First submitted 2025-01-05; First posted 2025-01-10 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Non Hodgkin Lymphoma
Keywords: refractory disease; chimeric antigen; B cell lymphomas; Cereblon E3 Ligase Modulators (CELMoD); immunomodulatory drugs (IMiD); tumor microenvironment (TME)
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Disease; Lymphoma, B-Cell | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Escalation of golcadomide combined with nivolumab at standard dosing will follow a standard 3+3 design with sequential cohorts of 3 participants. The first cohort will be treated at the 0.2 mg (14 days) dose level.
  Dose levels for Golcadomide:
  * Dose level 0: 0.1 mg (14 days)
  * Dose level 1: 0.2 mg (14 days) (starting dose)
  * Dose level 2: 0.4 mg (14 days)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- GOLCADOMIDE + Nivolumab 480 mg IV (Experimental): GOLCADOMIDE PO QD (Day 1-14) Nivolumab 480 mg IV (Q4 wk)
  Continue up to 24 cycles or until intolerable toxicity or disease progression
  Interventions: Drug: GOLCADOMIDE; Drug: Nivolumab

INTERVENTIONS:
Drug: GOLCADOMIDE — Golcadomide (GOLCA, CC-99282) is an oral cereblon E3 ligase modulator (CELMoD®) agent with immunomodulatory and tumor cell-autonomous activities. It is a modulator of the E3 ubiquitin ligase complex containing cereblon (CRL4-CRBN E3 ubiquitin ligase), with potential immunomodulating and antineoplastic activities.
  Other Names: Golcadomide (GOLCA; CC-99282)
Drug: Nivolumab — Nivolumab is an immune checkpoint inhibitor targeted therapy drug that blocks the PD-1 (programmed death receptor-1) pathway to help prevent cancer cells from hiding from the immune system, boosting the immune system's response.

SUMMARY:
In this combined phase I/II, open label, single arm trial to study, the safety and efficacy of combination Golcadomide and nivolumab in patients with non-Hodgkin lymphoma (NHL) who have experienced refractory/residual disease, at or after 30 days of receiving chimeric antigen T-cell (CAR-T) therapy will be studied. A dose escalation phase will be followed by a dose expansion design.

DETAILED DESCRIPTION:
Non-Hodgkin lymphoma (NHL) is a diverse group of lymphoid neoplasms affecting 80,470 new cases in the USA every year.1 Among the common types of NHL, diffuse large B-cell lymphoma (DLBCL) carries a five-year survival of 64.4% (SEER). Prognosis depends on disease specific factors such as stage and extent of spread, in addition to patient specific factors, such as age and performance status. Prior studies suggest that anti-PD-1 therapy may be effective in this population, especially if there is a way to further sensitize tumor cells to anti-PD-1 therapy to reduce T-cell exhaustion and increase inflammatory cytokines. Exposure to CELMoDs in addition to anti-PD1 therapy following CAR-T relapse may lead to deeper and more durable responses through re-expansion of CAR-T cells and modulation of tumor microenvironment (TME). This trial hypothesizes that combination Golcadomide at the selected dose and nivolumab at standard dosing will be safe and effective and that an overall response rate 45% or greater with a maximum dose-limiting toxicity (DLT) rate of 25% would be sufficient to warrant further interest in this combination in patients who have refractory NHL after 30 days of receiving therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed informed consent and willingness to comply with all study requirements for the duration of the study.
2. Patients 18 years of age or older.
3. Patients must have histologically confirmed high-grade large B-cell lymphoma such as diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL grade 3B), primary mediastinal B-cell lymphoma (PMBCL). Patient with transformation from indolent to large cell lymphoma will be allowed to enroll in the study.
4. Presence of FDG avid, radiographically measurable disease (Deauville 4-5) per Lugano 2014 response criteria which will include patients with metabolic partial response (PR), stable disease (SD), and progressive disease (PD), as assessed by the investigator.
5. Patients who received FDA-approved CD19-directed CAR T-cell product(s) (exclusive of any investigational CAR T-cell products).
6. Evidence of measurable residual disease 30 days and up to 1 year after receiving CAR-T therapy. Screening visit should be performed no later than day 365 after CAR-T infusion.
7. Eastern Cooperative Oncology group ECOG performance status ≤ 2.
8. Patients must have adequate organ and marrow function as defined in the protocol at the time of consent. Abnormalities reasonably attributed to underlying lymphoma will be allowed (e.g. anemia due to marrow involvement or LFT elevation due to metastatic involvement)
9. Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load are eligible.
10. For patients with evidence of chronic hepatitis virus infection (HBV or HCV), the viral load must be undetectable on suppressive therapy, if indicated.
11. Patients with CNS relapse (as an extension of systemic disease) are eligible, as determined by the investigator.
12. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. The malignancy should not be progressing or requiring active systemic treatment within the past year.
13. Patients with known history or current symptoms of cardiac disease should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification and may require an echocardiogram at the discretion of the investigator. To be eligible for this trial, patients should be class II, stage B or better.
14. Females of childbearing potential (FCBP) must have a negative pregnancy test during screening.
15. All subjects of childbearing potential must agree to use contraceptive methods (hormonal or barrier method of birth control; abstinence) for the duration of the study and for at least 28 days after the last dose of golcadomide. Should a woman become pregnant while she or her partner is participating in this study, she should inform her treating physician and discontinue therapy immediately. Pregnancies (both those of female patients and female partners of male patients) are reported in the same manner as SAEs within 24 hours of the Investigator's knowledge.
16. Ability to take oral medication and be willing to adhere to the golcadomide and nivolumab regimen.

Exclusion Criteria:

1. Treatment with any intervening anti-cancer therapies (other than palliative radiation) following CAR-T therapy. This study is intended to be the first treatment of residual disease after CAR-T therapy.
2. Patients who have not recovered from AEs (other than hematologic) of prior anti-neoplastic therapy (i.e., have residual toxicities > Grade 1) for the exception of alopecia, that require active management.
3. Hypersensitivity reaction to any of the study drugs or their derivatives.
4. Medical or psychiatric co-morbidities that in the opinion of the treating physician may compromise either compliance with or tolerance of study drugs.
5. Patients with GI malabsorption that may compromise absorption of oral golcadomide.
6. Presence of active autoimmune disease.
7. Patients requiring strong CYP3A inducers or inhibitors will be excluded. Note:

   1. Avoid coadministration of moderate CYP3A inhibitors and
   2. Avoid coadministration of moderate CYP3A inducers until more information regarding the potential DDI risk is available.

   Patients previously taking strong CYP3A inhibitors/inducers will require a washout period of at least 14 days or 5 half-lives, whichever is shorter, prior to the initiation of study treatment.
8. Currently breastfeeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) / Recommended Phase 2 dose (RP2D) | Up to 56 days from start of treatment
  The number and type of Dose Limiting Toxicities experienced during the first two cycles of treatment will be observed and assessed (per NCI-CTCAE v5.0) to determine the Maximum tolerated dose (MTD) / recommended phase 2 dose (RP2D) of golcadomide combined with standard dose nivolumab in participants with NHL who experienced disease progression or relapse after receiving CAR-T therapy as determined.
Lugano Response Evaluation | Up to 36 months
  Occurrence of partial response or better (objective response) per the Lugano PET-CT treatment response criteria. The Lugano classification (2014) is a lymphoma staging system that includes response based on CT evaluation. Scoring: (1)=no uptake or no residual uptake (when used interim), (2)=slight uptake, but below blood pool (mediastinum), (3)=uptake above mediastinal, but below or equal to uptake in the liver, (4)=uptake slightly to moderately higher than liver, (5)=markedly increased uptake or any new lesion (on response evaluation). Complete metabolic response (CMR) (score of 1, 2 or 3 in nodal or extranodal sites with or without a residual mass. Partial metabolic response (PMR) (score of 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size), or stable disease or no metabolic response (score of 4 or 5 with no obvious change in FDG uptake)

SECONDARY OUTCOMES:
Adverse Events and Serious Adverse Events (Phase l - Dose Escalation) | Up to 56 days from start of treatment
  Incidence of severity of adverse events and serious adverse events at least possibly related to trial treatment, per NCI-CTCAE v5.0.
Adverse Events and Serious Adverse Events (Phase ll - Dose Expansion) | Up to 36 months
  Incidence of severity of adverse events and serious adverse events at least possibly related to trial treatment, per NCI-CTCAE v5.0.
Preliminary Efficacy per Lugano Response Evaluation | Up to 26 months
  Occurrence of partial response or better (objective response) per the Lugano PET-CT treatment response criteria. The Lugano classification (2014) is a lymphoma staging system that includes response based on CT evaluation. Scoring: (1)=no uptake or no residual uptake (when used interim), (2)=slight uptake, but below blood pool (mediastinum), (3)=uptake above mediastinal, but below or equal to uptake in the liver, (4)=uptake slightly to moderately higher than liver, (5)=markedly increased uptake or any new lesion (on response evaluation). Complete metabolic response (CMR) (score of 1, 2 or 3 in nodal or extranodal sites with or without a residual mass. Partial metabolic response (PMR) (score of 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size), or stable disease or no metabolic response (score of 4 or 5 with no obvious change in FDG uptake)
Progression-free survival (PFS) | Up to 36 months
  Median time patients do not experience disease progression per Lugano classification (2014). Lugano criteria is a staging system including CT response evaluation. Scoring: (1)=no uptake or no residual uptake (when used interim),(2)=slight uptake, but below blood pool (mediastinum),(3)=uptake above mediastinal, but below or equal to uptake in the liver,(4)=uptake slightly to moderately higher than liver,(5)=markedly increased uptake or any new lesion (on response evaluation). Disease progression score=4 or 5 in any lesion with an increase in intensity of FDG uptake from baseline (and/or new FDG-avid foci consistent with lymphoma). Complete metabolic response (CMR) (score=1, 2 or 3 in nodal or extranodal sites with or without a residual mass, partial metabolic response (PMR) (score= 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size), or stable disease or no metabolic response (score=4 or 5 with no obvious change in FDG uptake)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Galanina, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No